CLINICAL TRIAL: NCT04089020
Title: Psychosocial Supports for Walking to School Paired With a Walking School Bus
Brief Title: Walking to School Supports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other); University of Kansas (Other)
Responsible Party: Principal Investigator, Jordan Carlson, PhD, Doctoral Research Faculty, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000851
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2022-10

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosocial intervention (Experimental): Text messaging and health coaching over the telephone to address goal setting, monitoring, motivation, problem solving, and related skills, delivered over 6 weeks.
  Interventions: Behavioral: Support for walking to school

INTERVENTIONS:
Behavioral: Support for walking to school — 5 modules that address psychosocial skills, with ongoing text messaging.

SUMMARY:
This pilot study will test the feasibility and acceptability of an enhanced individual-level intervention delivered to 4th-6th graders to increase rates of walking to/from school. Up to 8 youth who do not already walk to school will be enrolled into the intervention. The theoretically-based intervention content will be delivered over 6 weeks through family-based telephone coaching sessions, ongoing short message service (SMS) text messaging, and activities and content on the study website.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children enrolled at Benjamin Banneker school
* Parents/child dyads who completed the Phase 1 survey OR respond to recruitment attempts and express interest in walking to school. Included parent/child dyads will be:

Those who do not participate in LINC program both before and after school 4+ days per week (child); Those who live within the school boundary and south of Meyer Blvd (i.e., close enough to an existing walking school bus route) or are willing to drop off and/or pick up the child at a place along an existing walking school bus route (i.e., remote drop off).

Exclusion Criteria:

* Children not enrolled at Benjamin Banneker school
* Those who participate in LINC program both before and after school 4+ days per week (child); Those who do not live within the school boundary and south of Meyer Blvd (i.e., close enough to an existing walking school bus route) or are not willing to drop off and/or pick up the child at a place along an existing walking school bus route (i.e., remote drop off).
* We will exclude each of the following special populations:

Adults unable to consent Prisoners Wards of the state Pregnant women may be included, but only in such capacity as parents of other children enrolled at Benjamin Banneker school

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Carlson, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
De-identified information may be available upon request.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psychosocial Intervention
Started | 32 (18 youth participants 14 parent participants)
Completed | 31 (18 youth participants 13 parent participants)
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: This study included parent/child dyads, however no data was collected at baseline for parents.
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention: "Satisfaction Questionnaire"
Description: Acceptability and preferences related to intervention content will be measured using a questionnaire developed for this study ("satisfaction questionnaire"). Families (both parent and child responding together) will respond to 5 items asking about satisfaction with the intervention components. Items are rated on a 10-pt scale (minimum:1- maximum:10), with higher values indicating greater satisfaction. They will respond to two additional open-ended questions asking which aspects of the intervention they liked most and least. These qualitative items will be summarized.
Time Frame: at 6 weeks, immediately after completion of the intervention
Population: The satisfaction questionnaire was completed by the families (parent and child responding together). Of the 14 participant families, 13 were successfully contacted to complete the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 13
score on a scale
  Did you like the text messages? | 9.83 (0.58)
  How did you like the materials? | 9.33 (1.0)
  How did you like the calls? | 9.33 (1.16)
  How did you like the program overall? | 9.82 (0.6)

2. Secondary Outcome: Frequency of Walking to School
Description: Number of walking trips to/from school per week (0 to 10) will be assessed using a daily (Mon-Fri) tracking questionnaire completed through RedCap.
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: walking trips
Arm/Group | Psychosocial Intervention
Number analyzed (Participants) | 18
walking trips | 4.10 (2.15)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Adverse events were only monitored for child participants.
Arm/Group | Psychosocial Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT04089020/Prot_SAP_000.pdf